CLINICAL TRIAL: NCT03102320
Title: Phase 1b Multi-indication Study of Anetumab Ravtansine (BAY94-9343) in Patients With Mesothelin Expressing Advanced or Recurrent Malignancies
Brief Title: Phase 1b Multi-indication Study of Anetumab Ravtansine in Mesothelin Expressing Advanced Solid Tumors
Acronym: ARCS-Multi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: ImmunoGen, Inc. (Industry); MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15834; 2016-004002-33 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Neoplasms
Keywords: cholangiocarcinoma; pancreatic cancer; triple-negative breast cancer; non-small cell lung cancer; thymic carcinoma; gastric including gastroesophageal junction cancer
MeSH Terms: conditions — Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Thymoma | interventions — Cisplatin; Gemcitabine; anetumab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cholangiocarcinoma (Experimental): Safety lead-in phase will determine the MTD of anetumab ravtansine administered in combination with cisplatin. Please note the study is no longer recruiting for the cholangiocarcinoma safety lead-in phase.
  During the main study phase anetumab ravtansine will be administered at the determined MTD in combination with cisplatin. Please note the main study phase for cholangiocarcinoma will no longer be going ahead.
  Interventions: Drug: Cisplatin; Drug: Anetumab ravtansine (BAY94-9343)
- Adenocarcinoma of the pancreas (Experimental): Safety lead-in phase will determine the MTD of anetumab ravtansine administered in combination with gemcitabine During the main study phase, anetumab ravtansine will be administered at the determined MTD in combination with gemcitabine
  Interventions: Drug: Gemcitabine; Drug: Anetumab ravtansine (BAY94-9343)
- Other solid tumors (Experimental): (Non-small cell adenocarcinoma of the lung (NSCLC adenocarcinoma), Adenocarcinoma of the breast - triple negative (TNBC), Gastric adenocarcinoma including gastroesophageal junction (GEJ Cancer, Thymic carcinoma) During the main study phase, anetumab ravtansine will be administered at dose of 6.5 mg/kg in solid tumors
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 25 mg/m2 IV administered on day 1 and day 8 of 21 day cycle, for up to maximum 6 cycles
  Arms: Cholangiocarcinoma
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV administered on days 1 and 8 of a 21-day cycle
  Arms: Adenocarcinoma of the pancreas
Drug: Anetumab ravtansine (BAY94-9343) — Anetumab ravtansine 6.5mg/kg IV in monotherapy indications. For combination indications, the MTD determined in safety lead in phase will be administered

SUMMARY:
The key purpose of the main part of the study is to assess efficacy and safety of anetumab ravtansine as monotherapy or combination therapy for mesothelin expressing advanced solid tumors.

The main purpose of the safety lead-in (dose-finding) part of the study is to determine the safety and tolerability of anetumab ravtansine in combination with cisplatin and in combination with gemcitabine, and to determine the MTD of anetumab ravtansine in combination with cisplatin for mesothelin expressing advanced cholangiocarcinoma and in combination with gemcitabine for mesothelin expressing advanced adenocarcinoma of the pancreas.

Patients will receive anetumab ravtansine every three weeks in monotherapy for most indications. In cholangiocarinoma and adenocarinoma of the pancreas, 3-weekly anetumab ravtansine is administered in combination with cisplatin or gemcitabine respectively (both administered in a 2 week on / 1 week off schedule).

Treatment will continue until disease progression or until another criterion for withdrawal is met. .Efficacy will be measured by evaluating the tumor's objective response rate. Radiological tumor assessments will be performed at defined time points until the patient's disease progresses.

Blood samples will be collected for safety, pharmacokinetic and biomarker analysis. Archival or fresh biopsy tissue will also be collected for mesothelin expression testing and biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

* Availability of tumor tissue for mesothelin expression testing and for further biomarker analysis
* Histologically-confirmed, mesothelin-expressing metastatic or advanced non-metastatic disease (tumour type specific inclusion criteria)
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (or for thymic carcinoma, at least one measurable lesion per International Thymic Malignancy Interest Group (ITMIG) modified RECIST 1.1 criteria
* Adequate bone marrow, liver, renal and coagulation function
* Left ventricular ejection fraction (LVEF) ≥ 50% of the lower limit of normal (LLN) according to local institutional ranges
* Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Exposure to more than one prior anti-tubulin/microtubule agent
* Corneal epitheliopathy or any eye disorder that may predispose the patients to this condition
* Symptomatic Central nervous system (CNS) metastases and/or carcinomatous meningitis
* Contraindication to both CT and MRI contrast agents
* Active hepatitis B or C infection
* Pregnant or breast-feeding patients
* Tumor type specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Number of patients in the safety lead-in (SLI) phase who completed Cycle 1 or had a DLT and were not replaced. | At least 3 weeks after the last patient starts treatment
  During SLI, patients with cholangiocarcinoma received anetumab ravtansine in combination with cisplatin and patients with pancreatic adenocarcinoma received anetumab ravtansine in combination with gemcitabine. The highest dose of anetumab ravtansine that can be given so that not more than 1 out of 6 patients experiences a dose-limiting toxicity (DLT) during the DLT evaluation period were declared as the MTD for anetumab ravtansine in combination with cisplatin or with gemcitabine.
Objective response (qualitative improvement from baseline) of anetumab ravtansine for monotherapy and combination therapy in mesothelin expressing advanced solid tumors | Up to approximately 26 months after patient starts treatment
  A patient is a responder if the patient has a best response compared to baseline of complete response (CR) or partial response (PR) among all post-baseline tumor assessments, as determined per RECIST 1.1 criteria (ITMIG modified RECIST 1.1 criteria for thymic carcinoma)
Durable disease control (lack of progression from baseline) of anetumab ravtansine in indications pancreatic and gastric cancer (co-primary endpoint) | Up to approximately 26 months after patient starts treatment
  A patient experiences durable disease control if the patient has a tumor response compared to baseline of CR, PR or stable disease (SD) among the post-baseline tumor assessments made at least 180 days from first treatment, without prior disease progression

SECONDARY OUTCOMES:
Number of serious and non-serious adverse events (AEs) | Approximately 26 months (Until 30 days after the last day of study treatment, or until later resolution of adverse events or determination by the investigator that the event will not improve)
  Include treatment-emergent AEs, SAEs, treatment-related AEs, AEs of special interest, and deaths.
Disease control rate (DCR) | Up to approximately 24 months after last patient starts treatment, or until earlier disease progression [assessed every 6 weeks for the first 6 months, every 9 weeks until end of year 1 and every 12 weeks thereafter]
  The DCR is defined as the number of patients with disease control divided by the number of treated patients.
Duration of response (DOR) | Up to approximately 24 months after last patient starts treatment, or until earlier disease progression [assessed every 6 weeks for the first 6 months, every 9 weeks until end of year 1 and every 12 weeks thereafter]
  DOR is defined in responders as the time from documentation of tumor response (CR or PR) to earlier of disease progression or death
Durable response rate (DRR) | Up to approximately 24 months after last patient starts treatment, or until earlier disease progression [assessed every 6 weeks for the first 6 months, every 9 weeks until end of year 1 and every 12 weeks thereafter]
  A durable responder is defined as a responder (CR or PR) with a duration of response per RECIST 1.1 criteria (ITMIG modified RECIST 1.1 criteria for thymic carcinoma) of 180 days or more. The DRR is the number of durable responders divided by the number of treated patients.
Progression free survival (PFS) | Up to approximately 24 months after last patient starts treatment, or until earlier disease progression [assessed every 6 weeks for the first 6 months, every 9 weeks until end of year 1 and every 12 weeks thereafter]
  PFS is defined as time from start of treatment until disease progression according to RECIST 1.1 (ITMIG modified RECIST 1.1 criteria for thymic carcinoma) or death.
Durable disease control rate (DDCR) of anetumab ravtansine in indications other than pancreatic and gastric cancer | Up to approximately 24 months after last patient starts treatment, or until earlier disease progression [assessed every 6 weeks for the first 6 months, every 9 weeks until end of year 1 and every 12 weeks thereafter]
  A patient experiences durable disease control if the patient has a tumor response of CR, PR or SD with CR, PR or SD assessed at least 180 days from first treatment, without prior progression.

CONTACTS AND LOCATIONS:
Locations (72):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford Health Care, Stanford, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - National Cancer Institute - Maryland, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute, Farmington Hills, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, PA, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (8):
  - Blacktown Cancer & Haematology Centre, Blacktown, New South Wales
  - Mid North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Epworth HealthCare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Healthcare, Subiaco, Western Australia
- Belgium (4):
  - Hôpital Erasme/Erasmus Ziekenhuis, Bruxelles - Brussel
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre - UHN, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- France (12):
  - Hopital Jean Minjoz, Besançon
  - Hôpital Henri Mondor, Créteil
  - Centre Oscar Lambret - Lille, Lille
  - Centre Léon Bérard, Lyon
  - C.H.U. Timone, Marseille
  - Centre René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Centre Eugène Marquis - Rennes Cedex, Rennes
  - Institut Gustave Roussy, Villejuif
- Italy (6):
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - A.O.U. di Modena - Policlinico, Modena, Emilia-Romagna
  - Istituto Clinico Humanitas - Humanitas Mirasole S.p.A., Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - A.O.U.I. Verona, Verona, Veneto
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Maastricht UMC, Maastricht
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Universitario Quirón de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital del Mar, Barcelona
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón | Oncología, Madrid
  - Hospital Ramón y Cajal | Oncología, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Virgen de la Victoria, Málaga
- Switzerland (2):
  - Ospedale Regionale Bellinzona, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
- United Kingdom (6):
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Belfast City Hospital, Belfast, North Ireland
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Guy's Hospital, London
  - Royal Marsden Hospital (London), London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.